CLINICAL TRIAL: NCT00887393
Title: Effect of Macrocomposition on Nonalcoholic Fatty Liver Disease (NAFLD) in Bariatric Surgery Candidates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Elif Oral, Assoc. Prof. Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCRU 2462
Record Dates: First submitted 2009-04-22; First posted 2009-04-24 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Morbid Obesity; Non-alcoholic Fatty Liver Disease
Keywords: morbid obesity; non-alcoholic fatty liver disease; bariatric surgery; low fat diet; low carbohydrate diet
MeSH Terms: conditions — Obesity, Morbid; Non-alcoholic Fatty Liver Disease | interventions — Diet, Carbohydrate-Restricted; Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low carbohydrate (Other): Low carbohydrate pre-bariatric surgery diet
  Interventions: Other: low carbohydrate diet
- Low fat (Other): Low fat pre-bariatric surgery diet
  Interventions: Other: low-fat diet

INTERVENTIONS:
Other: low carbohydrate diet — 1000 to 1200 kcalorie low carbohydrate diet (< 15% of total kcaloric intake)
  Arms: Low carbohydrate
Other: low-fat diet — 1000 to 1200 kcalorie low-fat diet (30% fat, 60% carbohydrates of total kcaloric intake)
  Arms: Low fat

SUMMARY:
Nonalcoholic Liver disease (NAFLD) is known to be caused by deposition of fat in the liver. The impact of NAFLD on bariatric surgery is of great concern. Enlarged fatty livers increase the operative complications of bariatric surgery and weight loss prior to bariatric surgery has been shown to reduce complications of surgery. Most bariatric surgery programs use a conventional low fat, calorie restricted diet during the preparation phase for surgery. The investigators will compare the effects of the low carbohydrate versus the low fat diets on weight loss, reduction in liver fat content, and liver size. These results will provide new clinical insights into the optimal dietary intervention to make bariatric surgery safe and effective for the increasing numbers of patients opting for this aggressive therapy for morbid obesity. Patients approved for bariatric surgery by the University of Michigan Bariatric Surgery multidisciplinary committee will be randomly assigned to either a 1000 to 1200 calorie low fat or low carbohydrate, 8-week study diet. All the food for this study will be provided for free by the study team. Participants will be required to meet with the study team weekly to pick up study food and for a nutritional consult. These visits will occur in the eight weeks preceding the patient's bariatric surgery procedure. During the bariatric surgery, a liver biopsy will be performed to assess the impact of the study diet on liver fat content.

DETAILED DESCRIPTION:
The obesity epidemic has lead to increased morbidity and morality from cardiovascular disease and Type 2 diabetes. One co-morbidity of obesity is nonalcoholic fatty liver disease (NAFLD), which is characterized by excess fat deposition in the liver. About a third of the overweight and obese population has NAFLD and this rises to 80 to 90% of morbidity in obese patients. Short-term weight loss and caloric restriction leads to a reduction in hepatic fat content, suggesting an ability of the liver to quickly respond to dietary interventions. Manipulation of the diet macronutrient composition in order to achieve quicker weight loss as well as improve adverse metabolic consequences attributable to excess weight has attracted much attention and controversy. Multiple clinical studies have shown that low carbohydrate diets can provide more rapid weight loss in individuals in the short-term and that most have no trouble adhering to the diet for up to 6 months. Most bariatric surgery programs use a conventional low fat, calorie restricted diet during the preparation phase for surgery. However, no systematic comparison of diets with different macronutrient compositions have been performed. In this study we propose to compare the clinical effects of a low carbohydrate versus a low fat diet in individuals which can derive an immediate benefit from interventions that have the potential to reduce hepatic fat content: individuals that are preparing for bariatric surgery (laparoscopic Roux-en-Y gastric bypass surgery or adjustable laparoscopic gastric banding). Enlarged steatotic livers increase the operative risk of bariatric surgery and weight loss prior to bariatric surgery has been shown to reduce operative risk. We hypothesize that the use of a 1000 to 1200 kcalorie low carbohydrate diet (< 15% of total kcaloric intake) during the preparation phase for bariatric surgery will cause a greater reduction in weight, hepatic fat content and hepatic volume compared to a "conventional" 1000 to 1200 kcalorie low-fat diet (30% fat, 60% carbohydrates of total kcaloric intake) and offer clinical advantages by making the technical aspects of surgery easier. Thus, the data collected will provide significant new clinical insights into the effect of diets with different macronutrient composition. These results will provide a basis for larger clinical trials to identify the optimal dietary intervention to make bariatric surgery safe and effective for the increasing numbers of patients opting for this aggressive therapy for morbid obesity.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be deemed as appropriate candidates by the University of Michigan Bariatric Surgery multidisciplinary committee to undergo laparoscopic Roux-Y gastric bypass surgery or adjustable laparoscopic banding surgery
* Age 18 to 65 years
* Willing and able to give informed consent
* Clinical diagnosis of non-alcoholic fatty liver disease based on presence of abnormal LFTS and/or abnormal liver ultrasound
* Able to have an MRI procedure (able to fit into scanner, largest width < 60 cm, weight < 400 lbs, largest girth < 74 inches, do not have a pacemaker, artificial limbs or any other medical devices that contain iron that may be affected by the MRI procedure).
* Willing and able to tolerate the MRI procedure (use of benzodiazepines to complete the procedure is allowed if needed and deemed safe by the study team)

Exclusion Criteria:

* Clinical history of diabetes or fasting glucose > 126 mg/dl
* Alcohol consumption of > 40 grams/week
* Any other liver disease
* BMI < 40 kg/m2
* Unable to ambulate
* Any other factor that in the opinion of the PI or co-investigators which may impede successful completion of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2009-04; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of a low carbohydrate vs. a conventional low fat diet to reduce hepatic steatosis | 8-9 weeks
Compare differences in weight loss with a 2 month hypocaloric conventional low fat vs. low carbohydrate diets in individuals who are candidates for laparoscopic Roux-en-Y gastric bypass surgery or adjustable laparoscopic banding surgery | 8-9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elif A Oral, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States